CLINICAL TRIAL: NCT00447226
Title: A Phase II, Placebo Controlled, Double-Blind, Randomized, Discontinuation Study of Lapatinib Administered Orally to Subjects With ErbB2 Positive Ovarian, Gastric/Esophageal Adenocarcinoma, Uterine Serous Papillary, or Bladder Cancer
Brief Title: Randomized Discontinuation Study of Lapatinib Versus Placebo in Subjects With Documented Tumor Progression After Chemotherapy, or Where no Approved Therapy Exists
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study had failed to meet the primary objective of tumor response rate at 12 weeks from first dose.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LPT108741
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Cancer
Keywords: Ovarian Cancer; Bladder Cancer; ErbB2 positive; Lapatinib; Gastric/Esophageal Cancer; Uterine Serous Papillary Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapatinib Oral Tablets (Experimental)
  Interventions: Drug: Oral lapatinib tablets or placebo tablets
- Placebo Control (Placebo Comparator)
  Interventions: Drug: Oral lapatinib tablets or placebo tablets

INTERVENTIONS:
Drug: Oral lapatinib tablets or placebo tablets — Subjects administered open label lapatinib, 1500 mg to be taken orally once a day, for 12 weeks. After 12 weeks, subjects with a partial or complete response per Response Evaluation Criteria in Solid Tumors (RECIST) will continue to receive open label lapatinib (1500 mg/day orally) until disease progression. Subjects who maintain stable disease will be randomized in a 1:1 ratio to enter stage 2 of the study and receive double blind therapy of either lapatinib 1500 mg/day orally or placebo. Subjects who progress on placebo will have the option to receive lapatinib 1500 mg/day orally until further progression. Those who progress on lapatinib will be withdrawn from the study.

SUMMARY:
This study will examine the efficacy and safety of lapatinib in patients with ErbB2 positive ovarian, gastric/esophageal adenocarcinoma, uterine serous papillary, or bladder cancers.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age >= 18 years old.
* Life expectancy of at least 12 weeks.
* Have histologically confirmed ovarian, gastric/esophageal adenocarcinoma, uterine serous papillary, or bladder cancer.
* Have ErbB2-positive cancer as determined by Fluorescence In Situ Hybridization (FISH) assay.
* Have documented tumor progression after receiving all standard/approved chemotherapies per National Comprehensive Cancer Network (NCCN) guidelines (V1) for their specific cancer and no approved therapy exists.
* Have one or more tumors measurable by medical imaging and assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Have archived tumor tissue available for biomarker analysis.
* Have a negative serum pregnancy test if female of childbearing potential.
* Any chemotherapy, major surgery, or irradiation must have been completed at least 3 weeks prior to receiving study drug (6 weeks for mitomycin-C or nitrosourea) and subject must have recovered from all toxicities incurred as a result of previous therapy.
* Have a gastrointestinal tract intact enough to swallow and assure absorption of the drug.
* Women of childbearing potential must have a negative serum pregnancy test at screening and must use an approved contraceptive method, if appropriate (for example, intrauterine device, birth control pills, or barrier device) beginning 2 weeks before the first dose of investigational product and for 28 days after the final dose of investigational product. Males able to father a child must practice adequate methods of birth control or practice complete abstinence from intercourse from the first dose of investigational treatment until one week after the final dose of investigational treatment.
* Have a cardiac ejection fraction within institutional range of normal as measured by either echocardiogram or multigated acquisition scans. The same method of cardiac evaluation must be used consistently throughout the study.
* Subjects must have adequate organ function:

Hematologic:

absolute neutrophil count >1.5 x 109/L hemoglobin >9 g/dL platelets >75 x 109/L

Hepatic:

albumin >2.5 g/dL serum bilirubin <1.25 x upper limit of normal aspartate aminotransferase/alanine aminotransferase <3 x ULN if no documented liver metastases aspartate aminotransferase/alanine aminotransferase <5 x ULN with documented liver metastases

Renal:

serum creatinine <2.0 mg/dL

* OR - calculated creatinine clearance1 >40 mL/min

Exclusion Criteria:

* Have New York Heart Association Class III or IV, cardiac disease, myocardial infarction within past 6 months, unstable arrhythmia or evidence of ischemia on electrocardiogram.
* Subjects who have had chemotherapy or radiotherapy within 3 weeks prior to entering the study or who have unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment.
* Concurrent treatment with an investigational agent or participation in another treatment clinical trial.
* Prior lapatinib therapy.
* ECOG Performance Status 2 or greater.
* Subjects receiving concurrent chemotherapy, radiation therapy, immunotherapy, biologic therapy (including an ErbB1 and/or ErbB2 inhibitor), or hormonal therapy for treatment of their cancer. Concurrent treatment with bisphosphonates is allowed.
* History of allergic reactions attributed to compounds of similar chemical composition (quinazolines) to lapatinib.
* Concurrent treatment with prohibited medications.
* Malabsorption syndrome, resection of the small bowel or active, uncontrolled ulcerative colitis.
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety.
* Uncontrolled infection.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (20):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Leesburg, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Vancouver, Washington

REFERENCES:
- [Derived] Galsky MD, Von Hoff DD, Neubauer M, Anderson T, Fleming M, Nagarwala Y, Mahoney JM, Midwinter D, Vocila L, Zaks TZ. Target-specific, histology-independent, randomized discontinuation study of lapatinib in patients with HER2-amplified solid tumors. Invest New Drugs. 2012 Apr;30(2):695-701. doi: 10.1007/s10637-010-9541-0. Epub 2010 Sep 22. PMID 20857170

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants maintaining stable disease (SD) in Stage 1 (open label) were randomized to double-blind lapatinib 1500 milligrams (mg)/day or placebo (Stage 2). Of 32 participants in Stage 1, 7 maintained SD and were randomized into Stage 2. These 7 participants are represented as "completed" in the "Open-label Phase" participant flow table.
Groups:
- Placebo: Identical matching placebo orally, once a day
- Lapatinib 1500 Milligrams (mg): Lapatinib 1500 mg orally, once a day
Period: 12-Week Open-label Phase
Arm/Group | Placebo | Lapatinib 1500 Milligrams (mg)
Started | 0 | 32
Completed | 0 | 7
Not Completed | 0 | 25
Not completed — Adverse Event | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Disease Progression | 0 | 20
Not completed — Physician Decision | 0 | 1
Period: Double-blind Phase
Arm/Group | Placebo | Lapatinib 1500 Milligrams (mg)
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Disease Progression | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants treated in the open-label phase (1500 milligrams [mg] lapatinib, orally once a day), including those subsequently randomized to lapatinib (1500 mg, orally once a day) or matching placebo
Arm/Group | All Participants
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31
  African American/ African heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Tumor Response at 12 Weeks From First Dose
Description: Per Response Evaluation Criteria In Solid Tumors (RECIST): Complete response (CR), disappearance of all lesions; partial response (PR), >=30% decrease in the measurements of the largest lesions; stable disease (SD), insufficient shrinkage to qualify for PR or insufficient increase to qualify for progressive disease (PD); PD, >=20% increase in measurements of lesions or appearance of new lesions. Data were not fully analyzed due to early study termination.
Time Frame: Week 12
Population: All treated: all participants who received at least one dose of open-label lapatinib.
Measure: Number; unit: participants
Groups:
- Open-label Lapatinib 1500 Milligrams (mg): Open-label lapatinib 1500 mg orally, once a day
Arm/Group | Open-label Lapatinib 1500 Milligrams (mg)
Number analyzed (Participants) | 32
participants
  Complete response | 1
  Partial response | 0
  Stable disease | 9
  Progressive disease | 20
  Unknown | 2

2. Primary Outcome: Percentage of Participants Who Remained Progression-free 12 Weeks After Randomization
Description: The percentage of participants who did not show signs of progressive disease 12 weeks after receiving lapatinib or placebo in Stage 2 of the study (participants who maintained SD in Stage 1 were randomized to either lapatinib or placebo) was measured. Formal statistics for treatment comparison were not performed, due to early study termination. The percentage of participants displayed below includes those with CR + PR + SD.
Time Frame: Week 12 after randomization.
Population: Intent-to-Treat Population: all participants randomized to study treatment in Stage 2
Measure: Number; unit: percentage of participants
Groups:
- Double-blind Lapatinib 1500 mg: Double-blind lapatinib 1500 mg orally, once a day
Arm/Group | Double-blind Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 3 | 4
percentage of participants | 0 | 25

3. Secondary Outcome: Duration of Response
Description: Duration of response was calculated as the time from first documented partial response (PR; >=30% decrease in the measurements of the largest lesions) or complete response (CR; disappearance of all lesions) until disease progression, the time when the participant began a new anti-cancer therapy, or death. Data were not analyzed due to early study termination.
Time Frame: (assessments every 12 weeks until death for withdrawn participants and every 3 weeks for participants continuing on lapatinib)
Population: All treated: all participants who received at least one dose of open-label lapatinib.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Open-label Lapatinib 1500 mg: Open-label lapatinib 1500 mg orally, once a day
Arm/Group | Open-label Lapatinib 1500 mg | Double-blind Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was calculated as the time from the start of treatment until disease progression or death. For participants who did not have disease progression or did not die, the date on which alternative anti-cancer therapy began was used, or the date of last contact (if sooner). The word used for such participants was "censored". Data were not analyzed due to early study termination.
Time Frame: From start of treatment to disease progression/death (assessments every 12 weeks until death for withdrawn participants and every 3 weeks for participants continuing on lapatinib)
Population: All treated: all participants who received at least one dose of open-label lapatinib.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Open-label Lapatinib 1500 mg | Double-blind Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Time to Disease Progression (TTP)
Description: Time to disease progression was calculated as the time from the start of treatment to disease progression or death due to disease progression. For participants who did not progress, the date of last contact was used and for those who died due to other causes, the date of death was used. The word used for such participants was "censored". As the median value in the placebo arm was not reached (2 participants were censored and 2 were ongoing), results for the placebo arm are not displayed in the table below.
Time Frame: From start of treatment to disease progression/death (up to 83.3 weeks)
Population: All Treated: all participants who received at least one dose of open-label lapatinib.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Open-label Lapatinib 1500 mg: Open-label lapatinib 1500 mg orally, once a day: up to end of Stage 1
- Double-blind Lapatinib 1500 mg: Double-blind lapatinib 1500 mg orally, once a day: up to end of Stage 2
- Placebo: Identical matching placebo orally, once a day: up to end of Stage 2
Arm/Group | Open-label Lapatinib 1500 mg | Double-blind Lapatinib 1500 mg | Placebo
Number analyzed (Participants) | 32 | 3 | 0
weeks | 78 [42 to 92] | 137 [41 to 164] |

6. Secondary Outcome: Number of Participants With the Indicated Change in Cancer Antigen-125 (CA-125) Levels From Day 1
Description: CA-125 is a "tumor marker", found in greater concentration in tumor cells than other cells of the body. In particular, CA-125 is present in greater concentration in ovarian cancer cells than in other cells. A decreasing level generally indicates that therapy has been effective, whereas an increasing level indicates tumor recurrence.
Time Frame: Pre-dose and every 6 weeks until withdrawal (up to 84.1 weeks)
Population: Participants with ovarian cancer. The number of participants for whom there are data varies at each time point, depending on how many participants had CA-125 samples.
Measure: Number; unit: participants
Groups:
- All Participants With Ovarian Cancer: All participants with ovarian cancer treated in the open-label phase (1500 mg lapatinib, orally once a day), including those subsequently randomized to lapatinib (1500 mg, orally once a day) or matching placebo
Arm/Group | All Participants With Ovarian Cancer
Number analyzed (Participants) | 10
participants
  CA-125 doubled at Week 6, n=3 | 1
  CA-125 halved at Week 6, n=3 | 0
  CA-125 doubled at Week 18, n=2 | 0
  CA-125 halved at Week 18, n=2 | 0
  CA-125 doubled at withdrawal at <=12 weeks, n=4 | 3
  CA-125 halved at withdrawal at <=12 weeks, n=4 | 0
  CA-125 doubled at withdrawal at >12 weeks, n=1 | 0
  CA-125 halved at withdrawal at >12 weeks, n=1 | 0

7. Secondary Outcome: Incidence of MET Amplification in Gastric Cancer
Description: The number of gastric cancer participants with MET amplification (determined by fluorescence in situ hybridization [FISH] assay) compared to the total number of gastric cancer participants screened was to be recorded. Amplification of the MET gene has been reported to be related to carcinogenesis, progression of gastric cancer, and poor prognosis. Data were not analyzed due to early study termination.
Time Frame: Performed on archived tissue collected at screening.
Population: All participants with gastric cancer who were screened to determine their eligibility to enter into the study
Measure: Number; unit: participants per total screened
Groups:
- Screened Participants With Gastric Cancer: Screened participants with gastric cancer
Arm/Group | Screened Participants With Gastric Cancer
Number analyzed (Participants) | 0

8. Secondary Outcome: Incidence of ErbB2-positive Participants
Description: The number of ErbB2-positive participants (determined by FISH assay) compared to the total number of participants screened was to be recorded. Over-expression of ErbB2 has been correlated with an overall poor prognosis. Data were not analyzed, due to early study termination.
Time Frame: Screening
Population: All participants who were screened to determine their eligibility to enter into the study
Measure: Number; unit: participants per total screened
Groups:
- All Screened Participants: All screened participants
Arm/Group | All Screened Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and serious adverse events (SAEs), regardless of relationship to lapatinib, were collected from the first dose until 5 days after the last dose of study medications (up to 84.1 weeks).
Description: The AEs and SAEs presented below represent data collected from all participants, whether taking open-label lapatinib or whether randomized to lapatinib/placebo. The SAE of cerebral hemorrhage was reported 2 days after the last dose of study drug was taken and was thus not an "on-treatment" event.
Groups:
- All Participants: All participants treated in the open-label phase (1500 mg lapatinib, orally once a day), including those subsequently randomized to lapatinib (1500 mg, orally once a day) or matching placebo
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 4/32
Other Adverse Events (participants affected / at risk) | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=32)
Ataxia (Nervous system disorders) | 1
Cerebral hemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Cellulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=32)
Diarrhea (Gastrointestinal disorders) | 17
Fatigue (General disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Edema peripheral (General disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Anemia (Blood and lymphatic system disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Insomnia (Psychiatric disorders) | 4
Pyrexia (General disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Weight decreased (Investigations) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Failure to thrive (Metabolism and nutrition disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Cellulitis (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Mucosal inflammation (General disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Infections and infestations) | 2
Pollakiuria (Renal and urinary disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin chapped (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Urinary tract infection (Infections and infestations) | 2

LIMITATIONS AND CAVEATS:
Study terminated prematurely: preliminary assessment (prompted by low screening/enrollment rates) showed primary objective of tumor response rate not met. Also unable to test primary treatment comparison after randomization following SD at 12 wks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.